CLINICAL TRIAL: NCT02089399
Title: An Open Label, Randomized, 2-Sequence, Multiple-Dose, Cross-Over Study to Investigate the Drug-Drug Interaction of Sevikar and Crestor in Healthy Adult Volunteers
Brief Title: Pharmacokinetics and Drug Interaction Study Between Amlodipine,Olmesartan and Rosuvastatin in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DW_DWJ1351001
Record Dates: First submitted 2014-03-14; First posted 2014-03-17 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
MeSH Terms: interventions — olmesartan; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment AB (Experimental): S->S+C
  Interventions: Drug: Sevikar(amlodipne/olmesartan); Drug: crestor(Rosuvastatin)
- Treatment C (Experimental): C
  Interventions: Drug: crestor(Rosuvastatin)

INTERVENTIONS:
Drug: Sevikar(amlodipne/olmesartan) — Treatment AB
  Arms: Treatment AB
Drug: crestor(Rosuvastatin) — Treatment AB/Treatment C

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics profile and drug-drug interaction between amlodipine, olmesartan and rosuvastatin in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 19 - 55 years
* A body mass index in the range 19 - 27 kg/m2
* Willingness to participate during the entire study period
* Written informed consent after being fully informed about the study procedures

Exclusion Criteria:

* Any past medical history of hepatic, renal, gastrointestinal, respiratory, endocrine, psychiatric, neurologic, haemato-oncologic or cardiovascular disease
* History of clinically significant drug hypersensitivity
* Use of medication within 7 days before the first dose
* Heavy drinker (>140 g/week)
* Whole blood donation during 60 days before the study
* Judged not eligible for study participation by investigator

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
AUCtau | Multiple blood sample will be collected for 24 hours after last dosing in each of the treatment
Css,max | Multiple blood sample will be collected for 24 hours after last dosing in each of the treatment

SECONDARY OUTCOMES:
Tss,max | Multiple blood sample will be collected for 24 hours after last dosing in each of the treatment
Css,min | Multiple blood sample will be collected for 24 hours after last dosing in each of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea